CLINICAL TRIAL: NCT04935814
Title: Cardiac Output Response to Vasopressin Infusion In Abdominal Surgery Patients Under Mechanical Ventilation: A Clinical Pharmacodynamics Study
Brief Title: Cardiac Output Response to Vasopressin Infusion In Abdominal Surgery Patients Under Mechanical Ventilation
Acronym: CORVaso
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CORVaso / RBHP 2021 GODET 2
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Major Abdominal Surgery; General Anesthesia; Mechanical Ventilation; Vasopressin Infusion
Keywords: Vasopressin; Argipressin; Cardiac Output; General Anesthesia; Mechanical Ventilation
MeSH Terms: conditions — Diabetes Insipidus | interventions — Arginine Vasopressin

STUDY DESIGN:
Intervention Model Description: CORVaso is a pharmacological trial which aims to determine the variations of cardiac output during vasopressin infusion in major abdominal surgery patients.
Masking Description: Patients are under general anesthesia and outcomes assessor (statistician) will be blinded of patients positions orders.
  Sequential positions of patients will be randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous vasopressin infusion (Experimental): After general anesthesia, patients will receive a continuous infusion of vasopressin in order to improve mean arterial pressure by 20 mmHg.
  Interventions: Drug: Vasopressin, Arginine

INTERVENTIONS:
Drug: Vasopressin, Arginine — Once vasopressin infusion started, patients positions will be randomized: Trendelenburg (-30°), anti Trendelenburg (+30°) and supine position (0°).

SUMMARY:
In this study, the investigators propose to explore the hemodynamic variations induced by vasopressin and its influence on cardiac output, mean systemic pressure, and venous return resistance measured through cardiopulmonary interactions, according to the approach proposed by Guyton, in patients undergoing major abdominal surgeries.

DETAILED DESCRIPTION:
Maintaining hemodynamic stability is one of the main objectives of the anesthesiologist or the intensivist, either in the ICU or the OR. This consists of optimizing cardiac output to ensure satisfactory systemic perfusion during the peri-operative period or the ICU stay. The occurrence of oxygen debt (mismatch between oxygen consumption and transport) and/or tissue hypoperfusion are key factors in the development of organ failure. Numerous studies have shown in recent years that individualized hemodynamic optimization (cardiac output and organ perfusion pressure) reduces the risk of postoperative and ICU morbidity and mortality.

Monitoring of cardiac output and stroke volume is a valuable and essential aid in determining the therapies to be used for this optimization, whether it involves volume expansion or the use of a vasopressor or even inotropic agent.

Several vasopressor therapies have been available to date. Norepinephrine is currently the reference in the treatment of vasoplegic shock states, but also in the operating room during major surgery or in fragile patients. Other molecules are currently available and are used in a disparate manner, according to the habits of each practitioner, sometimes outside regulatory rules, not following international recommendations concerning the pathology in question: adrenaline, dopamine, phenylephrine, terlipressin...

Vasopressin (D-arginine-D-vasopressin) is an endogenous hormone synthesized by the hypothalamus (peptide composed of 9 amino acids) which has an antidiuretic renal action through its V2 receptor but also a vasoconstriction activity through its V1a receptor, at the level of the smooth muscles of the vascular wall. It also participates in the stimulation of catecholamine secretion by the adrenal medulla. Vasopressin is commercially available under the name "argipressin". It is currently indicated as an adjunct to other vasopressors such as norepinephrine in refractory septic shock to maintain satisfactory hemodynamic stability.

However, its vasoconstrictive and hemodynamic effects, including its influence on cardiac output, have never been studied to date and to the knowledge of investigators. In particular, there are no studies showing the influence of this molecule on mean systemic pressure and venous return resistance, which are fundamental determinants of its impact on left heart function and thus on cardiac output.

In this study, the investigators propose to explore the hemodynamic variations induced by vasopressin and its influence on cardiac output, mean systemic pressure, and venous return resistance measured through cardiopulmonary interactions, according to the approach proposed by Guyton.

ELIGIBILITY:
Inclusion Criteria:

* Adults above 18
* Planned for a major abdominal surgery under general anesthesia
* Under mechanical ventilation
* Presence of a central venous and arterial lines allowing transpulmonary thermodilution cardiac output measurement
* Patient's consent with a social insurance

Exclusion Criteria:

* Do not consent to participate
* History of heart attack, arteriopathy or aneurysm
* Contraindication to use transpulmonary thermodilution to measure cardiac output :
* coagulopathy
* cardiac arrythmia
* presence of pace-maker or defibrillator
* severe valvulopathy
* Patients with Acute Respiratory Distress Syndrome (according to Berlin criteria)
* History of arterial hypertension (treated or not)
* History of seizure, chronic headache, asthma or heart failure
* Left Ventricular Ejection Fraction (LVEF) < 45% or right ventricular dysfunction
* History of pulmonary lobectomy or surgery
* History of restrictive or obstructive pulmonary disease
* Body Mass Index (BMI) < 15 or > 40 kg/m²
* Pregnancy
* Known allergy to vasopressin
* Patients under protection of justice (guardianship, curators...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Variation of cardiac output after an infusion of vasopressin at different levels of cardiac preload | 15 minutes after position change
  Using a thermodilution method, cardiac output will be measured and recorded at different levels of cardiac preload obtained by changing patient's position (Trendelenburg, anti-Trendelenburg and supine position).

SECONDARY OUTCOMES:
Variation of mean systemic filling pressure and venous return after an infusion of vasopressin at different levels of cardiac preload | 15 minutes after position change
  Mean systemic filling pressure will be determined by plotting the venous return curve using the cardiopulmonary interaction described by Guyton, by changing patient's position (Trendelenburg, anti-Trendelenburg and supine position).
Variation of central venous pressure after an infusion of vasopressin at different levels of cardiac preload | 15 minutes after position change
  Using a central venous catheter, the central venous pressure will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Godet, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France